CLINICAL TRIAL: NCT07068399
Title: Use of Shock Wave Therapy for Neo-Vascularisation in Non-critical Coronary Artery Disease: Validation by Quantitative Cardiac MRI Perfusion
Acronym: CSWT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UW 19-651
Record Dates: First submitted 2025-07-07; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-02

CONDITIONS: Coronary Artery Disease
Keywords: Stress Cardiac Magnetic Resonance; Cardiac Extracorporeal Shock Wave Therapy
MeSH Terms: conditions — Coronary Artery Disease | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CSWT (Experimental): Cardiac patients who have progressively increasing coronary plaque burden that is not yet at a critical stage of the CAD process and are randomised to the group receiving extracorporeal shock wave therapy. Cardiac MRI scans will be done before the treatment and 6 months after the end of CSWT.
  Interventions: Procedure: Extracorporeal shock wave therapy
- No intervention (No Intervention): The other half of similar cardiac patients who do not receive CSWT. Optimised medical therapy will be given to patients in this group. Cardiac MRI scans will be done twice.

INTERVENTIONS:
Procedure: Extracorporeal shock wave therapy — Extracorporeal shock wave therapy (ESWT) delivers acoustic energy transmitted through liquid medium to internal body tissues. The intervention group will receive a total of 9 ESWT treatment sessions and 200 shocks will be applied to each ischaemic zone of myocardium for 3 times a week on the three weeks that the patients receive ESWT.
  Other Names: CSWT; Cardiac ESWT
  Arms: CSWT

SUMMARY:
This is a randomised controlled trial aimed to demonstrate the effect of cardiac extracorporeal shock wave therapy (CSWT) on the angiogenesis effect of myocardium by determining myocardial perfusion and left ventricular function in patients with coronary artery disease (CAD) when measured by cardiac MRI before and after the treatment.

DETAILED DESCRIPTION:
In 2017 a systematic review of extracorporeal shock wave therapy (ESWT) in the treatment of coronary artery disease was undertaken by Berneikaite G. et al. to perform meta-analysis regarding anti-anginal efficacy of Cardiac ESWT (CSWT). The review identified 39 studies encompassing 1,189 patients with 1006 patients treated by CSWT. The meta-analysis found all selected studies demonstrated significant improvement in subjective measures of angina symptoms and/or quality of life, while the majority of studies also found improvement in left ventricular function and myocardial perfusion. For myocardial perfusion, SPECT was employed in 27 of 32 studies and PET in 2 of 4 studies. Cassar et al compared myocardial segments that were treated with CSWT and those segments that were not, finding after 4 months of follow-up that the progression of Ischaemic burden of untreated segments was significantly greater. As Cardiac MRI has not been employed to monitor myocardial perfusion in these studies, and with the increasing number of reports demonstrating the usefulness of MRI in characterising ischaemia, it seems opportune to utilise this non-radioactive technology to study the beneficial effect of CSWT in non-critical Coronary artery cases who have been found to have serially increasing coronary plaque burden. It has been shown that efficacious Statin usage can progressively regress coronary plaque volume, so augmenting collateral flow at stenotic coronary sites would buy time for Statin usage to complete this regression for definitive cure of CAD. With the availability of MRI methods to quantify myocardial perfusion accurately, the efficacy of CSWT for Neovascularization can thus be effectively documented as numerical data using Quantitative Cardiac MRI Perfusion, accompanied by Bull's eye views for ease of visual appreciation.

ELIGIBILITY:
Inclusion criteria:

* Patients with symptoms of coronary artery disease
* Patients without obstructive coronary artery disease
* with LVEF not < 40%.

Exclusion criteria:

* Age < 18 years,
* Pregnancy or lactation.
* Contraindication to contrast enhanced stress Cardiac Magnetic Resonance (eg. Estimated GFR <30ml/min/1.73m2, severe allergy to gadolinium based contrast agent, contraindication to adenosine)
* Life expectancy <24 months
* Haemodynamically unstable
* Participation in other clinical trial within 6 months of enrollment.
* Recent myocardial infarction within 6 months.
* Unable to consent to or perform components of the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Myocardial perfusion | 6 months and 3 weeks
  Quantitative magnetic resonance imaging with resting and and stress perfusion imaging will be performed.

SECONDARY OUTCOMES:
Left ventricular function | 6 months and 3 weeks
  Quantitative magnetic resonance imaging with resting and and stress perfusion imaging will be performed

CONTACTS AND LOCATIONS:
Locations (1):
- HKU Li Ka Shing Faculty of Medicine, Hong Kong, Hong Kong